CLINICAL TRIAL: NCT02221544
Title: The Effect of Low-frequency Repetitive Transcranial Magnetic Stimulation on Motor Function in Patients With Parkinson's Disease (PD) With Freezing of Gait (FOG).
Brief Title: The Effect of Low-frequency rTMS on Motor Function in PD Patients With Freezing of Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director of the R&D division in the Tel Aviv Sourasky Medical Center (TASMC), Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-13-NG-599-CTIL
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, rTMS, Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS treatment followed by Sham (Experimental): A course of low-frequency repetitive transcranial magnetic stimulation (rTMS) delivered over the supplementary motor area (SMA) followed by rTMS maintenance period (1 month) and followed by sham treatment in order to show the efficacy of treatment
  Interventions: Device: Low-frequency repetitive Transcranial Magnetic Stimulation; Device: rTMS maintenance; Device: Sham; Device: Sham maintenance
- Sham treatment followed by rTMS (Experimental): A course of sham followed by followed by sham maintenance period (1 month) and than followed by low-frequency repetitive transcranial magnetic stimulation (rTMS) delivered over the supplementary motor area (SMA) in order to show the effectiveness of rTMS
  Interventions: Device: Low-frequency repetitive Transcranial Magnetic Stimulation; Device: rTMS maintenance; Device: Sham; Device: Sham maintenance

INTERVENTIONS:
Device: Low-frequency repetitive Transcranial Magnetic Stimulation — Participants will receive treatment at a frequency of 3 sessions per week for 4 weeks (12 sessions). In each session patient will receive repetitive Transcranial Magnetic Stimulation using a stimulation frequency of 10 Hz for half an hour.
  The treatment is done by attaching an electromagnetic coil to the scalp using a special hat. Each patient has a personal hat which serves him throughout the entire process. The treatment is performed without anesthesia and patient fully conscious. During the treatment he sits comfortably on a chair, meanwhile the magnetic field passes through the skull into the brain.
  Other Names: rTMS treatment
Device: rTMS maintenance — Same treatment as in rTMS treatment intervention, but only once a week for a month
Device: Sham — Participants will receive sham treatment at a frequency of 3 sessions per week for 4 weeks (12 sessions total) for half an hour each session. The treatment is done by attaching an electromagnetic coil to the scalp but without turning on the magnetic field.
Device: Sham maintenance — The same as Sham stimuli intervention, but once a week for a month

SUMMARY:
This study is a double blind comparative study examining the effectiveness of the rTMS treatment on Freezing of Gait (FOG) phenomenon in patients with Parkinson's disease. We hypothesize that treatment using rTMS stimulation on frontal lobe areas will improve gait quality and decrease the frequency of FOG in patients with Parkinson's disease.

DETAILED DESCRIPTION:
A course of low-frequency repetitive transcranial magnetic stimulation (rTMS) delivered over the supplementary motor area (SMA) improves motor symptoms in patients with Parkinson's disease (PD).

The present study is a comparative study that examines the effectiveness of rTMS treatment technique Freezing of Gait (FOG) phenomenon in Parkinson's disease patients. We hypothesize that treatment using rTMS stimulation on frontal areas will decreasing frequency of FOGs in patients with Parkinson's disease and improve gait quality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease (PD), as diagnosed by a neurologist.
2. The mini-mental state examination questionnaire score above 24 points.
3. Suffer from a disabling phenomenon called Freezing of Gait (FoG) (Freezing Of Gait questionnaire score> = 10)
4. Negative responses to the Preliminary Safety Magnetic Stimulation Treatment questionnaire.

Exclusion Criteria:

1. Other neurological or psychiatric disorders.
2. Severe personality disorder.
3. High Blood Pressure.
4. History of epilepsy, seizures or convulsions.
5. History of epilepsy or convulsions in first-degree relatives.
6. History of head injury or stroke.
7. Metal remains of the skull or inside the brain (outside the oral cavity).
8. Surgeries including metallic implants or known history of metal particles in the eye, pacemakers, hearing devices transplantation, or medical pumps.
9. Current history of migraines for the last six months.
10. A history of drug or alcohol abuse
11. Other medical research in the time to experiment or three months ahead. -

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency and severity of the freezing of gait phenomenon | One week post intervention
  The new version of the Freezing of Gait questionnaire will be used to quantify the frequency and severity of this symptom. The score will be compared to baseline.

SECONDARY OUTCOMES:
Community ambulation | One week post intervention
  Will be assessed using 1) the Habitual Physical Activity Questionnaire (HPAQ). It will quantify the type and amount of regular physical activity. 2) A body-worn small lightweight device that will be worn by the subject for 7 days to monitor stepping and physical activity.
Changes in endurance | One week post intervention
  This measure will be assessed using the 2 minute walk test. The distance walked during 2 minutes will be compared to baseline performance.
Balance | One week post intervention
  Balance and lower extremity function will be assessed using performance-based measures: (1) The Four Square Step Test (FSST), (2) The Short Physical Performance Battery (SPPB), and (3) The Mini- Balance Evaluation Systems Test (mini-BEST).
Immediate changes in blood pressure | Every session, immediately after receiving the treatment
  Measuring blood pressure will monitor subjects' autonomic response to the treatment. Measures will be compared before and after receiving the treatment
Immediate change in gait function | One week post intervention
  Gait speed and variability will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel